CLINICAL TRIAL: NCT02033681
Title: Optimal Time Delay of Epinephrine Injection With "One-per-mil" Tumescent Solution to Visualize Operation Field in Hand Surgery Without Tourniquet
Brief Title: Optimal Time Delay of Epinephrine Injection With "One-per-mil" Tumescent Solution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Theddeus O. H. Prasetyono, Research Coordinator of Plastic Surgery Division, Faculty of Medicine, University of Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPM-1
Record Dates: First submitted 2013-09-03; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Ischemia
Keywords: epinephrine; hand; ischemia; lidocaine; upper extremity
MeSH Terms: conditions — Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "One-per-mil" Tumescent Solution (Experimental)
  Interventions: Procedure: "One-per-mil" Tumescent Solution Injection
- Saline Solution (Placebo Comparator)
  Interventions: Procedure: Saline Solution

INTERVENTIONS:
Procedure: "One-per-mil" Tumescent Solution Injection — "One-per-mil" tumescent solution containing 1:1,000,000 epinephrine concentration in saline solution, is injected to the finger.
  Arms: "One-per-mil" Tumescent Solution
Procedure: Saline Solution — Saline solution is injected into the tissue as a placebo control.
  Arms: Saline Solution

SUMMARY:
The aim of this study is to know the characteristic of "one-per-mil" tumescent solution in regards of the optimal time delay to achieve optimal visualization of operation field in hand and digit surgery.

Hypothesis:

1. Epinephine in "one-per-mil" concentration by tumescent injection technique will provide faster decrease in oxygen saturation compared to normal saline solution injected by tumescent technique.
2. Epinephrine in "one-per-mil" concentration by tumescent injection technique will provide effectiveness in vasoconstriction longer than 10 minutes as the optimal time delay.
3. Epinephine in "one-per-mil" concentration by tumescent injection technique causes no finger necrosis as normal saline solution injected by tumescent technique.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind study to measure the optimal time delay of 1:1,000,000 epinephrine in saline solution injected by tumescent technique until maximum vasocontriction in the distal finger is achieved.

Subjects will be injected in both his ring fingers(distal phalanges, volar side) with randomized solutions, one containing "one-per-mil" tumescent solution and the other containing only normal saline solution; information which both the injector and examiner are blinded from. Maximum vasoconstriction of the finger injected is depicted by the lowest oxygen saturation (recorded every minute until 45 minutes using pulse oxymeter).

ELIGIBILITY:
Inclusion Criteria:

* Willing to join the research
* BMI 18.5-23
* Healthy individual, no history of blood or coagulation disorders

Exclusion Criteria:

* BMI <18.5 or >23
* History of blood or coagulation disorder, diabetes mellitus, heavy smoker

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Time to achieve lowest oxygen saturation | 45 minutes
  After being injected with the solution, the ring finger is put on a continuous monitoring of pulse oxymeter, while the examiner records the decrease of oxygen saturation every minute until 45 minutes length of time. The time when lowest oxygen saturation is achieved is recorded, depicting the optimal time delay to achieve maximum vasoconstriction of the finger after injection.

SECONDARY OUTCOMES:
Pain Sensation | 45 minutes
  Pain sensation of the finger's pulp was examined (using VAS) and recorded every 15 minutes. These data will be compared to the baseline data prior to injection.
Tactile Sensation | 45 minutes
  Tactile sensation of the finger's pulp was examined (using Semmes Weinstein Touch Test) and recorded every 15 minutes after the injection. We will compare this data with the baseline data collected prior to injection.
Complication | 6 hours
  Subjects will be observed for 6 hours after the injection to record any sign and symptoms related to the complication of the procedure (persisted pain, pallor, numbness).
Decrease in fingertip's temperature | 45 minutes
  After injection, temperature of fingertip is measured and recorded every 15 minutes for total time of 45 minutes. The data will be compared with baseline temperature recorded before injection

CONTACTS AND LOCATIONS:
Overall Officials: Theddeus OH Prasetyono, MD, Principal Investigator — Plastic Surgery Division, Faculty of Medicine University of Indonesia/Cipto Mangunkusumo Hospital
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia